CLINICAL TRIAL: NCT02187536
Title: Pharmacokinetics of Single Oral Doses of 40 mg Simvastatin and Its Metabolite Simvastatin Acid With and Without Concomitant Administration of Telmisartan 80 mg Daily, Given Orally Over 6 Days. A Randomised, Placebo Controlled, Double Blind (for Telmisartan), Two Way Cross Over Trial in Healthy Subjects
Brief Title: Pharmacokinetics of Simvastatin and Its Metabolite Simvastatin Acid With and Without Concomitant Administration of Telmisartan in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 502.341
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; Simvastatin

ARMS (2):
- Telmisartan combined with Simvastatin (Experimental): Telmisartan once daily (day 1 to day 6) and Simvastatin given once (day 6)
  Interventions: Drug: Telmisartan; Drug: Simvastatin
- Simvastatin and telmisartan placebo (Active Comparator): Telmisartan placebo once daily (day 1 to day 6) and Simvastatin given once (day 6)
  Interventions: Drug: Simvastatin; Drug: Telmisartan placebo

INTERVENTIONS:
Drug: Telmisartan
  Arms: Telmisartan combined with Simvastatin
Drug: Simvastatin
Drug: Telmisartan placebo
  Arms: Simvastatin and telmisartan placebo

SUMMARY:
To assess the pharmacokinetics of simvastatin and simvastatin acid with/without concomitant administration of telmisartan

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by results of screening
* Signed written informed consent in accordance with good clinical practice (GCP) and local legislation
* Age ≥ 18 and ≤ 55 years
* Broca ≥ -20 % and ≤ +20 %

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastro-intestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Supine blood pressure at screening of systolic ≤ 110 mmHg and diastolic ≤ 60 mmHg
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infection
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half life (> 24 hours) ≤ 1 month prior to administration or during the trial
* Use of any drugs which might influence the results of the trial (≤ 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (30 days prior to administration or during the trial)
* Smoker
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≤ 1 month prior to administration or during the trial)
* Excessive physical activities (≤ 5 days prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance
* Hypersensitivity to telmisartan and/or simvastatin and/or related classes of drugs

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (e.g. sterilization, intrauterine device (IUD), oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2000-04; Primary Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of simvastatin and simvastatin acid in plasma at different time points (AUC) | Pre-dose, up to day 32 after start of treatment
Maximum concentration of simvastatin and simvastatin acid in plasma (Cmax) | Pre-dose, up to day 32 after start of treatment

SECONDARY OUTCOMES:
Time to Cmax after a single extravascular dose (tmax) | Pre-dose, up to day 32 after start of treatment
Elimination half-life in plasma (t1/2) | Pre-dose, up to day 32 after start of treatment
Total clearance from plasma (CLtot/f) | Pre-dose, up to day 32 after start of treatment
Mean time of residence in the body (MRTtot) | Pre-dose, up to day 32 after start of treatment
Apparent volume of distribution during the terminal phase (Vz/f) | Pre-dose, up to day 32 after start of treatment
Area under the plasma concentration-time curve of telmisartan at steady state (AUCss) | Pre-dose, up to day 32 after start of treatment
Maximum concentration of telmisartan in plasma at steady state (Cmax,ss) | Pre-dose, up to day 32 after start of treatment
Number of patients with clinically relevant findings in laboratory values | Pre-dose, up to day 32 after start of treatment
Number of patients with clinically relevant findings in vital signs (blood pressure, pulse rate) | Pre-dose, up to day 32 after start of treatment
Number of patients with adverse events | Up to day 32 after start of treatment
Number of patients with clinically relevant findings in ECG | Pre-dose, up to day 32 after start of treatment